CLINICAL TRIAL: NCT05093491
Title: Ultrasonographic Evaluation of Respiratory Muscles in Stroke Patients and Correlation With Pulmonary Function Tests
Brief Title: Ultrasonographic Evaluation of Respiratory Muscles in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FTRTEZDOGAN
Record Dates: First submitted 2021-09-20; First posted 2021-10-26 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Muscle; Pulmonary Function Test
Keywords: stroke; pulmonary function; ultrasound; respiratory muscle thickness
MeSH Terms: conditions — Stroke | interventions — Spirometry; Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: Ultrasonographic measurements were performed of the bilateral diaphragm and abdominal muscle thickness and thickening ratio of stroke patients. Spirometry evaluation was performed by another investigator. Diagnostic Test: Bilaterally diaphragm and abdominal muscle thickness and thickening ratio with ultrasonography
  Interventions: Diagnostic Test: Spirometry and ultrasonography in stroke group
- Healthy individuals: Ultrasonographic measurements were performed of dominant side diaphragm and abdominal muscle thickness and thickening ratio. Spirometry evaluation was performed by another investigator. Diagnostic Test: Dominant side diaphragm and abdominal muscle thickness and thickening ratio with ultrasonography
  Interventions: Diagnostic Test: Spirometry and ultrasonography in healthy group

INTERVENTIONS:
Diagnostic Test: Spirometry and ultrasonography in stroke group — Ultrasonographic measurements were performed of the bilateral diaphragm and abdominal muscle thickness and thickening ratio in the supine position in the stroke patient group. The spirometric evaluation was also performed
  Groups: Stroke patients
Diagnostic Test: Spirometry and ultrasonography in healthy group — Ultrasonographic measurements were performed of dominant side diaphragm and abdominal muscle thickness and thickening ratio in the supine position in healthy individuals group. The spirometric evaluation was also performed
  Groups: Healthy individuals

SUMMARY:
Ultrasonographic evaluation of respiratory muscle thickness in stroke patients, determination of its correlation with pulmonary function test (PFT) , and the first evaluation method to determine respiratory rehabilitation goals and to use it in the follow-up of the effectiveness of the treatment.

DETAILED DESCRIPTION:
The study is planned as a cross-sectional prospective study. Healthy volunteers and stroke patients who are planned to be hospitalized in the Stroke clinic for rehabilitation in Istanbul Physical Medicine Rehabilitation Training and Research Hospital are evaluated and included in the study according to the inclusion and exclusion criteria.

Demographic data of patients (gender, age, height, weight, body mass index, comorbidity status, smoking/alcohol use, dominant extremity, stroke etiology, duration, side), functional status (Brunnstrom stages, Functional Ambulation Scale (FAS), Daily Living Activity (ADL) Index), Pulmonary Function Test (PFT) measurement results and bilateral diaphragm and abdominal muscle thicknesses and thickening ratio in ultrasonography, demographic data of healthy volunteers (gender, age, height, weight, body mass index, comorbidity status, smoking/alcohol use, dominant side), PFT measurement results and the dominant side diaphragm and abdominal muscle thicknesses and thickening ratio in ultrasonography is done and included in the study.

In the ultrasonographic evaluation of the participants, using a 7-12 Mhz linear Probe, measurements are made of the diaphragm at the end of tidal expiration and forced inspiration, abdominal muscles at the end of tidal expiration and at the end of forced expiration, while all respiratory muscles are lying in the supine position. Diaphragm thickness is measured between the 8th and 9th ribs at the level of the anteroaxillary line, rectus abdominis; 4 cm lateral of the umbilicus, transversus abdominis, external oblique, internal oblique muscles' measurement is made from the middle of the lowest part of the 12. rib and the highest point of the iliac crest and 2.5 cm in front of the midaxillary line. All measurements are repeated 3 times and the average value will be recorded.

Vital capacity[VC], forced vital capacity [FVC], forced expiratory volume 1 second [FEV1] , FEV1/FVC, maximal expiratory flow rate [PEF], maximum inspiratory pressure [MIP] maximum expiratory pressure [MEP] in patients' PFT ] measurement results are checked.

Intragroup and intergroup data are compared.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic or Hemorrhagic stroke patients
* Stroke duration >6 months
* Mini-mental test score >24

Exclusion Criteria:

* Individuals with acute or chronic lung disease
* Patients with a history of thoracic or abdominal surgery
* Patients with other neuromuscular diseases
* Aphasia type with impaired understanding
* Facial paralysis

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients and, healthy volunteers which have close demographic data with stroke patients
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2021-12-25 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Diaphragma and Abdominal Muscle Thickness and thickening ratio | 1 day (a single point in time)
  Diaphragma and Abdominal Muscle ultrasonographic millimetric measurement
Forced vital capacity [FVC] | 1 day (a single point in time)
  >%80 is normal results
Forced expiratory volume 1 second [FEV1] | 1 day (a single point in time)
  >%80 is normal results
FEV1/FVC | 1 day (a single point in time)
  >%80 is normal results
Maximal expiratory flow rate [PEF] | 1 day (a single point in time)
  >%80 is normal results
Maximum inspiratory pressure [MIP], | 1 day (a single point in time)
  >80cmH2O is normal results
Maximum expiratory pressure [MEP] | 1 day (a single point in time)
  >95cmH2O is normal results

SECONDARY OUTCOMES:
Brunnstrom stages | 1 day (a single point in time)
  min 1 max 6, bigger values mean better results,
Functional Ambulation Scale (FAS) | 1 day (a single point in time)
  min 0 max 5, bigger values mean better results,
Daily Living Activity (ADL) Index | 1 day (a single point in time)
  min 0 max 100, bigger values mean better results,

CONTACTS AND LOCATIONS:
Overall Officials: Yunus Emre Dogan, MD, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospita; Kadriye Ones, Prof, Study Chair — Istanbul Physical Medicine Rehabilitation Training and Research Hospita
Locations (1):
- Istanbul physical medicine rehabilitation training &research hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Misuri G, Colagrande S, Gorini M, Iandelli I, Mancini M, Duranti R, Scano G. In vivo ultrasound assessment of respiratory function of abdominal muscles in normal subjects. Eur Respir J. 1997 Dec;10(12):2861-7. doi: 10.1183/09031936.97.10122861. PMID 9493674
- [Result] Jung JH, Kim NS. The correlation between diaphragm thickness, diaphragmatic excursion, and pulmonary function in patients with chronic stroke. J Phys Ther Sci. 2017 Dec;29(12):2176-2179. doi: 10.1589/jpts.29.2176. Epub 2017 Dec 13. PMID 29643599
- [Result] Kim M, Lee K, Cho J, Lee W. Diaphragm Thickness and Inspiratory Muscle Functions in Chronic Stroke Patients. Med Sci Monit. 2017 Mar 11;23:1247-1253. doi: 10.12659/msm.900529. PMID 28284044
- [Result] Ishida H, Suehiro T, Kurozumi C, Ono K, Watanabe S. Correlation Between Abdominal Muscle Thickness and Maximal Expiratory Pressure. J Ultrasound Med. 2015 Nov;34(11):2001-5. doi: 10.7863/ultra.14.12006. Epub 2015 Sep 22. PMID 26396169